CLINICAL TRIAL: NCT01460472
Title: A Prospective, Randomized, Multicenter, Open Label Phase III Study of Active Specific Immunotherapy With Racotumomab Plus Best Support Treatment Versus Best Support Treatment in Patients With Advanced Non-small Cell Lung Camcer.
Brief Title: Immunotherapy With Racotumomab in Advanced Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Recombio SL (Industry)
Collaborators: CIMAB (Cuba) (Unknown); Laboratorio Elea Phoenix S.A. (Industry); Innogene Kalbiotech Pte. Ltd (Industry); Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-AR-1E10 MAb-301; ISRCTN47153584 (Registry Identifier: International Clinical Trials Register Platform (ICTRP), WHO)
Record Dates: First submitted 2011-10-23; First posted 2011-10-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: NSCLC; Lung Cancer, Non-small Cell
Keywords: NSCLC; Lung cancer, small-cell; advanced lung cancer; therapeutic vaccine; anti-idiotypic vaccine; 1E10
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — racotumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Racotumomab plus Best Support Treatment (Experimental): Patients will receive Racotumomab and Best Support Treatment, which includes any further onco-specific therapy for progressive disease.
  Interventions: Biological: Racotumomab
- Best Support Treatment (Active Comparator): Patients will receive best support treatment for advanced NSCLC including onco-specific therapies when disease progresses.
  Interventions: Other: Best Support Treatment

INTERVENTIONS:
Biological: Racotumomab — Patients will receive best support treatment and vaccination with racotumomab. The vaccination schedule is as follows: 5 doses (1mg/mL each), intradermally, every 2 weeks (induction period) followed by monthly vaccinations until any criteria for discontinuation are met. If disease progression occurs and further onco-specific therapy is indicated, the patient will be able to continue in the study and vaccination will not be interrupted unless criteria for vaccine discontinuation are met.
  Other Names: 1E10
  Arms: Racotumomab plus Best Support Treatment
Other: Best Support Treatment — Patients will receive best support treatment for advanced NSCLC as per each institution's standards, including onco-specific therapies when disease progresses.
  Arms: Best Support Treatment

SUMMARY:
This is a prospective, randomized, open label, parallel-group, multicenter phase III study to evaluate the efficacy and safety of active specific immunotherapy with racotumomab plus best supportive care versus best supportive care in patients with advanced NSCLC who have achieved an Objective Response (Partial or Complete Response) or Stable Disease with standard first-line treatment. Also immunological parameters will be evaluated. Best supportive therapy will be administered to all patients in the study according to institutional standards and includes any subsequent onco-specific therapies. 1082 patients will be included in the study, with non-small cell lung cancer in stages IIIA (non-resectable), IIIB or IV.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent.
2. Cytologic or histologically diagnosed NSCLC in stages IIIA (non-resectable) or IIIB or IV (TNM).
3. In continuous complete or partial remission or stable disease according to Response Evaluation Criteria in Solid Tumours (RECIST) after standard first-line treatment.
4. Imaging studies documenting the response to first-line therapy must be available for evaluation by the investigator.
5. Time lapse of 21 to 56 days between the end of onco-specific treatment and start of vaccination. Patients must have recovered from any acute toxicity produced by previous therapy.
6. Age greater than or equal to 18 years, either sex.
7. Eastern Cooperative Oncology Group performance status less than 2.
8. Adequate organ function, defined as follows:

   8.1. Electrocardiogram (ECG) without significant anomalies, performed in the 7 days preceding entry

   8.2. Haemoglobin greater than or equal to 90 g/L

   8.3. Total white blood cell count (WBC) greater than or equal to 3.0 x 10^9/L

   8.4. Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L

   8.5. Platelet count greater than 100 x 10^9/L

   8.6. Total bilirubin less than or equal to 1.5 fold the maximum normal value at the place of evaluation or 2.5 fold the maximum normal value in case of liver metastases

   8.7. Glutamic-oxaloacetic transaminase/aspartate aminotransferase (GOT/AST), and glutamic-pyruvic transaminase/alanine aminotransferase (GPT/ALT), less than or equal to 2.5 fold the maximum normal value at the place of evaluation (in case of liver metastasis, less than 5 fold the maximum normal value)

   8.8. Creatinine less than or equal to 2 mg/dL (less than or equal to 176 µmol/L)
9. Known hepatitis B virus carriers who have liver function tests within the accepted limits are eligible

Exclusion Criteria:

1. Pregnant or breastfeeding patients
2. Known hypersensitivity to any component of the formulation
3. Fertile patients of either sex who do not use adequate contraceptive methods while on treatment
4. Disease progression prior to randomization
5. Recurrent NSCLC, who relapse less than one year after completing curative intent therapy
6. Patients receiving other investigational medication (including investigational immunotherapy for NSCLC) or having received such medication within 30 days before entering the protocol
7. Autoimmune diseases or chronic decompensated diseases
8. Acute allergic disorders or a history of severe allergic reactions
9. Known brain metastases
10. History of demyelinating disease or inflammatory disease of the central nervous system or the peripheral nervous system
11. Non-controlled intercurrent diseases, including active infections, symptomatic congestive heart failure, unstable chest angina or heart arrhythmia, as well as mentally incapable patients
12. Other malignant diseases except non- melanoma skin cancer, in situ carcinoma of the cervix, incidental prostate cancer (T1a, Gleason less than or equal to 6, prostate specific antigen (PSA) less than 0.5 ng/ml) or any other tumour having received adequate treatment and evidencing a disease-free period greater than or equal to 5 years
13. Receiving chronic therapy for more than 10 days at doses of prednisone greater than 10 mg/day (or equivalent) at the moment of the inclusion. Inhaled and topical corticosteroids are allowed.
14. Active hepatitis C or positive tests for human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1082 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Until date of death or last censored observation, on average upto 17 months
  A comparison of survival in the subgroup of inoperable stage IIIA and dry IIIB will be performed in 757 (approximately 70% of the study population)

SECONDARY OUTCOMES:
Number of Participants with Adverse events as a measure of safety and tolerability | Until death, on average during 17 months
  Safety will be evaluated at each study visit according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 and will include physical examination with vital signs, performance status as per the Eastern Cooperative Oncology Group scale(ECOG scale), laboratory tests and clinical history.
Progression Free Survival | From randomization until date of first documented progression of disease, assessed as per RECIST 1.0 during an expected average of 17 months
  Tumour evaluations will be performed every 2 months and evaluated as per Response Evaluation Criteria in Solid Tumors (RECIST).
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside | Baseline
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside for Racotumomab Group | Month 3
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside for Racotumomab Group | Month 6
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside for Racotumomab Group | Month 9
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside for Racotumomab Group | Month 12
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside for Racotumomab Group | After the first year, every 3 months, on average for 17 months
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay. | Baseline
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay for Racotumomab Group. | Month 3
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay for Racotumomab Group. | Month 6
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay for Racotumomab Group. | Month 9
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay for Racotumomab Group. | Month 12
Evaluation of the reactivity if the antibodies against X63 tumor line (mouse myeloma) for Racotumomab Group | Baseline
Evaluation of the reactivity if the antibodies against X63 tumor line (mouse yeloma) for Racotumomab Group | Month 3
Evaluation of the reactivity if the antibodies against X63 tumor line (mouse myeloma) for Racotumomab Group | Month 6
Evaluation of the reactivity if the antibodies against X63 tumor line (mouse myeloma) for Racotumomab Group | Month 9
Evaluation of the reactivity if the antibodies against X63 tumor line (mouse myeloma) for Racotumomab Group | Month 12
Evaluation of the reactivity if the antibodies against X63 tumor line (mouse myeloma) for Best Support Treatment Group | Baseline
Evaluation of the reactivity if the antibodies against X63 tumor line (mouse myeloma) for Best Support Treatment Group | Month 4
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside for Best Support Treatment Group | Baseline
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside for Best Support Treatment Group | Month 4
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay for Best Support Treatment Group. | Month 4
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry. | Baseline
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry in the Racotumomab Group. | Month 3
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry in the Racotumomab Group. | Month 6
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry in the Racotumomab Group. | Month 9
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry in the Racotumomab Group. | Month 12
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry in the Best Support Treatment Group. | Month 4
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) | Baseline
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) in the Racotumomab Group. | Month 3
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) in the Racotumomab Group. | Month 6
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) in the Racotumomab Group. | Month 9
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) in the Racotumomab Group. | Month 12
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) in the Best Support Treatment Group. | Month 4
Measurement of pro-inflammatory and anti-inflammatory cytokines | Baseline
Measurement of pro-inflammatory and anti-inflammatory cytokines in the Racotumomab Group | Month 3
Measurement of pro-inflammatory and anti-inflammatory cytokines in the Racotumomab Group | Month 6
Measurement of pro-inflammatory and anti-inflammatory cytokines in the Racotumomab Group | Month 9
Measurement of pro-inflammatory and anti-inflammatory cytokines in the Racotumomab Group | Month 12
Measurement of pro-inflammatory and anti-inflammatory cytokines in the Best Support Treatment Group | Month 4
Determination of anti-idiotypic IgG response | Baseline
Determination of anti-idiotypic IgG response in the Racotumomab Group. | Month 3
Determination of anti-idiotypic IgG response in the Racotumomab Group. | Month 6
Determination of anti-idiotypic IgG response in the Racotumomab Group. | Month 9
Determination of anti-idiotypic IgG response in the Racotumomab Group. | Month 12
Determination of anti-idiotypic IgG response in the Best Support Treatment Group. | Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Gomez, M.D., Study Director — Recombio S.L.
Locations (46):
- Argentina (8):
  - Instituto Médico CER, Quilmes, Buenos Aires
  - Hospital Privado de Córdoba, Córdoba, Córdoba Province
  - Instituto Oncológico de Córdoba, Córdoba, Córdoba Province
  - Fundación COIR, Mendoza, Mendoza Province
  - ISIS Clinica Especializada, Santa Fe, Santa Fe Province
  - Policlínica Privada Instituto de Medicina Nuclear, Bahía Blanca
  - Hospital Italiano, Córdoba
  - Centro Oncológico de Rosario, Rosario
- Brazil (24):
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - NOB - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital Universitário de Brasília, Brasília, Federal District
  - Pro Onco - Centro de Tratamento Oncológico, Londrina, Paraná
  - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - UPCO - Unidade de Pesquisas Clínicas em Oncologia, Pelotas, Rio Grande do Sul
  - HCPA - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Universitário de Brasília, Brasília - DF
  - Centro de Oncologia do Parana, Curitiba
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza - CE
  - Hospital Amaral de Carvalho, Jaú
  - Pro Onco - Centro de Tratamento Oncológico, Londrina - PR
  - Centro Oncologico de Mogi das Cruzes, Mogi das Cruzes
  - Liga Norte Riograndense Contra o Cancer, Natal
  - Hospital da Cidade de Passo Fundo, Passo Fundo - RS
  - UPCO - Unidade de Pesquisas Clínicas em Oncologia, Pelotas - RS
  - Hospital Moinhos de Vento, Porto Alegre
  - HCPA - Hospital de Clínicas de Porto Alegre, Porto Alegre - RS
  - Oncologistas Associados, Rio de Janeiro
  - NOB - Nucleo de Oncologia da Bahia, Salvador - BA
  - Faculdade de Medicina do ABC, Santo André
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto
  - GRAM - Grupo de Assistencia Medica e Prestacao de Servicos, São Paulo
- Cuba (3):
  - Hospital "Hermanos Ameijeiras", Havana
  - Hospital "Celestino Hernández Robau", Provincia de Villa Clara
  - Hospital Jose Ramon Lopez Tabranes, Versalles
- Indonesia (5):
  - Dr Moewardi Hospital, Central Java
  - Persahabatan Hospital, Jakarta
  - RS Kanker 'Dharmais', Jakarta
  - Dr Soetomo Hospital, Surabaya
  - Dr Sardjito Hospital, Yogyakarta
- Philippines (2):
  - Perpetual Succour Hospital, Cebu City
  - Veterans Memorial Medical Center, Manila
- Johns Hopkins Singapore International Medical Centre, Singapore, Singapore
- Thailand (3):
  - Chiang Mai Hospital, Chiang Mai
  - Khon Kaen Hospital, Division of Pulmonary and Critical Care Medicine, Khon Kaen
  - Songklanagarind Hospital - HOCC-PSU, Songkhla